CLINICAL TRIAL: NCT03215979
Title: Use of Platelet-enriched Plasma to Improve the Percentage of Integration of the Cutaneous Graft During Second Stage of Auricular Reconstruction in Children Aged 8-12 Years; A Controlled Clinical Trial
Brief Title: Use of Platelet-enriched Plasma During Auricular Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Dr. Manuel Gea González (Other Government)
Responsible Party: Principal Investigator, Jorge Raúl Carrillo Córdova, Medical Doctor, Hospital General Dr. Manuel Gea González
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05-20-2017
Record Dates: First submitted 2017-07-07; First posted 2017-07-12 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Ear Cartilage; Platelets; Microtia-Anotia
MeSH Terms: conditions — Microtia-Anotia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP-Arm (Experimental): In this arm, surgeon will be applying platelet enriched plasma(PEP) (5 ml) during the second stage procedure of auricular reconstruction. PEP will be infected in the temporal fascia used to cover the cartilage frame.
  Interventions: Procedure: Platelet enriched plasma administration
- Placebo-Arm (Placebo Comparator): This arm will be used as control. The surgeon will inject 0.9% saline solution (5ml) in a blinded basis.
  Interventions: Procedure: Placebo Arm

INTERVENTIONS:
Procedure: Platelet enriched plasma administration — It is a blinded administration of platelet enriched plasma in the temporal fascia used to cover the auricular reconstruction frame, during the second stage of the procedure. The use of platelet enriched plasma is focused to improve the integration rate of the full-thickness split skin graft
  Arms: PEP-Arm
Procedure: Placebo Arm — 5 ml of saline 0.9%will be applied in the temporal fascia as a placebo used to compare to the experimental group.
  Arms: Placebo-Arm

SUMMARY:
In this study investigators are trying to determine the benefits of using platelet enriched plasma during the second stage of auricular reconstruction. The intervention will be blinded to the surgeon and the surgical team. The main outcome will be the evaluation of the integration rate of the skin full thickness graft used to coat the auricular frame.

ELIGIBILITY:
Inclusion Criteria:

* Microtia Tanzer II-A
* patients aged 8-12 years
* Haemoglobin > 10 gr/dL
* History of first stage of auricular reconstruction

Exclusion Criteria:

* associated endocrinopathies
* desnutrition (<2.5 gr/ dL)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-11-29 (Estimated); Study Completion 2018-12-10 (Estimated)

PRIMARY OUTCOMES:
Integration rate (in percentage) of the full thickness split graft sued during the second stage of auricular reconstruction. | evaluation will be at day 10
  Evaluation of the integration will be made on clinical basis, and evaluated by 3 experimented plastic surgeons.

SECONDARY OUTCOMES:
Complication | evaluation will be at day 10
  It refers to a deviation from the normal course of the pathology, 3 complications will be taken into account: infection, seroma and hematoma

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General "Dr. Manuel Gea González", Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No